CLINICAL TRIAL: NCT02575534
Title: Acute Mechanical Response to Anti-arrhythmic Drug Therapy
Acronym: AAD and CRT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment in study.
Sponsor: Evan Adelstein, MD (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Evan Adelstein, MD, Evan Adelstein, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO14010486
Record Dates: First submitted 2015-06-16; First posted 2015-10-14 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Arrhythmias
Keywords: anti-arrhythmic therapy
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Procainamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- observational (Experimental): All patients will undergo 12-lead ECG and transthoracic echocardiography on the day of the study. These studies will be performed on patients as their previously implanted device is reprogrammed to pace in different modes. Patients will then receive an infusion of procainamide (12 mg/kg up to a maximum of 1 g) at a rate of 20 mg/min. Repeat ECG and echocardiograms will then be performed.
  The patient's device will be programmed to a specific setting before and after the procainamide infusion.
  Interventions: Drug: Procainamide

INTERVENTIONS:
Drug: Procainamide — the procainamide will be infused at 12mcg/kg up to a max of 1 gram at a rate of 20mg/min which will take up to 1 hour to infuse
  Other Names: procan

SUMMARY:
The aim of this study is to determine if anti-arrhythmic drugs with a sodium channel-blocking mechanism exert a detrimental electromechanical effect on cardiac function in patients depending upon baseline intraventricular conduction and left ventricular function.

DETAILED DESCRIPTION:
Amiodarone therapy is used frequently for control of ventricular arrhythmias in patients who receive painful shocks from an implantable cardioverter-defibrillator (ICD). Data in post-myocardial infarction (MI) patients and ICD patients suggest that amiodarone is mortality-neutral; it neither confers increased nor decreased mortality. However, these data are derived from patients largely with normal intraventricular conduction, manifesting as a QRS complex duration on the surface ECG <120 ms. Amiodarone, in addition to potassium-channel blocking effects, is a sodium channel-blocker. Because sodium channels mediate cardiac depolarization, and a QRS complex >120 ms is indicative of abnormal depolarization, amiodarone may not be benign in patients with such conduction defects. Patients with cardiac resynchronization therapy-defibrillators (CRT-D), who all have abnormal baseline intraventricular conduction, may therefore be adversely affected by amiodarone. Anecdotal clinical data suggest that this may be the case, but the question of amiodarone's cardiac safety profile in CRT patients has never been studied.

ELIGIBILITY:
Inclusion Criteria:

* Implanted cardiac device requiring generator change and a new device
* Able to give informed consent

Exclusion Criteria:

* Current membrane-active anti-arrhythmic
* Glomerular filtration rate (GRF)<30 milliliters (mL)/min
* MAP<60 mmHg
* Known intolerance to procainamide
* Pregnancy
* Age <18 or >85 years old
* Baseline QT interval >480 ms (500 ms if paced)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Change in QRS duration | baseline and 1 hour post infusion
  the QRS waveform measurements will be calculated on the EKG prior to and after the procainamide infusion
changes in left ventricular volumes as measured via echocardiogram | baseline and 1 hour post infusion
  the left ventricular volume will be calculated via echocardiogram pre and post procainamide infusion
changes in ejection fraction as measured via echocardiogram | baseline and 1hour post infusion
  ejection fraction will be calculated via echocardiogram pre and post procainamide infusion.
changes in RV-LV electrical activation (in CRT patients) | baseline and 1 hour post infusion
  The RV-LV electrical activation will be assessed during the device interrogation pre and post procainamide infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Evan Adelstein, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Evan Adelstein, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Connolly SJ, Camm AJ, Halperin JL, Joyner C, Alings M, Amerena J, Atar D, Avezum A, Blomstrom P, Borggrefe M, Budaj A, Chen SA, Ching CK, Commerford P, Dans A, Davy JM, Delacretaz E, Di Pasquale G, Diaz R, Dorian P, Flaker G, Golitsyn S, Gonzalez-Hermosillo A, Granger CB, Heidbuchel H, Kautzner J, Kim JS, Lanas F, Lewis BS, Merino JL, Morillo C, Murin J, Narasimhan C, Paolasso E, Parkhomenko A, Peters NS, Sim KH, Stiles MK, Tanomsup S, Toivonen L, Tomcsanyi J, Torp-Pedersen C, Tse HF, Vardas P, Vinereanu D, Xavier D, Zhu J, Zhu JR, Baret-Cormel L, Weinling E, Staiger C, Yusuf S, Chrolavicius S, Afzal R, Hohnloser SH; PALLAS Investigators. Dronedarone in high-risk permanent atrial fibrillation. N Engl J Med. 2011 Dec 15;365(24):2268-76. doi: 10.1056/NEJMoa1109867. Epub 2011 Nov 14. PMID 22082198
- [Result] Packer DL, Prutkin JM, Hellkamp AS, Mitchell LB, Bernstein RC, Wood F, Boehmer JP, Carlson MD, Frantz RP, McNulty SE, Rogers JG, Anderson J, Johnson GW, Walsh MN, Poole JE, Mark DB, Lee KL, Bardy GH. Impact of implantable cardioverter-defibrillator, amiodarone, and placebo on the mode of death in stable patients with heart failure: analysis from the sudden cardiac death in heart failure trial. Circulation. 2009 Dec 1;120(22):2170-6. doi: 10.1161/CIRCULATIONAHA.109.853689. Epub 2009 Nov 16. PMID 19917887
- [Result] Echt DS, Liebson PR, Mitchell LB, Peters RW, Obias-Manno D, Barker AH, Arensberg D, Baker A, Friedman L, Greene HL, et al. Mortality and morbidity in patients receiving encainide, flecainide, or placebo. The Cardiac Arrhythmia Suppression Trial. N Engl J Med. 1991 Mar 21;324(12):781-8. doi: 10.1056/NEJM199103213241201. PMID 1900101
- [Result] Cardiac Arrhythmia Suppression Trial II Investigators. Effect of the antiarrhythmic agent moricizine on survival after myocardial infarction. N Engl J Med. 1992 Jul 23;327(4):227-33. doi: 10.1056/NEJM199207233270403. PMID 1377359
- [Result] Cairns JA, Connolly SJ, Roberts R, Gent M. Randomised trial of outcome after myocardial infarction in patients with frequent or repetitive ventricular premature depolarisations: CAMIAT. Canadian Amiodarone Myocardial Infarction Arrhythmia Trial Investigators. Lancet. 1997 Mar 8;349(9053):675-82. doi: 10.1016/s0140-6736(96)08171-8. PMID 9078198
- [Result] Julian DG, Camm AJ, Frangin G, Janse MJ, Munoz A, Schwartz PJ, Simon P. Randomised trial of effect of amiodarone on mortality in patients with left-ventricular dysfunction after recent myocardial infarction: EMIAT. European Myocardial Infarct Amiodarone Trial Investigators. Lancet. 1997 Mar 8;349(9053):667-74. doi: 10.1016/s0140-6736(96)09145-3. PMID 9078197
- [Result] Connolly SJ, Dorian P, Roberts RS, Gent M, Bailin S, Fain ES, Thorpe K, Champagne J, Talajic M, Coutu B, Gronefeld GC, Hohnloser SH; Optimal Pharmacological Therapy in Cardioverter Defibrillator Patients (OPTIC) Investigators. Comparison of beta-blockers, amiodarone plus beta-blockers, or sotalol for prevention of shocks from implantable cardioverter defibrillators: the OPTIC Study: a randomized trial. JAMA. 2006 Jan 11;295(2):165-71. doi: 10.1001/jama.295.2.165. PMID 16403928